CLINICAL TRIAL: NCT00903747
Title: A Phase I Thorough QT/QTc Study To Evaluate The Effect of Therapeutic and Supratherapeutic Multiple Doses of Prucalopride on Cardiac Repolarisation in Healthy Male and Female Volunteers
Brief Title: Thorough Corrected QT Interval (QTc) Study To Evaluate Possible Effects of Prucalopride on ECG Parameters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Remi Van Den Broeck, Movetis NV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0001-C102
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Constipation
Keywords: Prucalopride; safety study
MeSH Terms: conditions — Constipation | interventions — prucalopride; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prucalopride
  Interventions: Drug: prucalopride
- 2 (Placebo Comparator): Placebo/moxifloxacin
  Interventions: Drug: moxifloxacin; Drug: placebo

INTERVENTIONS:
Drug: prucalopride — 2-10 mg prucalopride
  Other Names: Resolor
  Arms: 1
Drug: moxifloxacin — 400 mg moxifloxacin (Group 2a)
  Other Names: Avelox
  Arms: 2
Drug: placebo — placebo (Group 2b)
  Arms: 2

SUMMARY:
This is a 2-arm, parallel-group active- and placebo-controlled, double-blind randomised study, stratified by gender and with a hybrid crossover group design, to compare treatment with prucalopride 2 mg/day (intended therapeutic dose) and prucalopride 10 mg/day (supratherapeutic dose) with placebo. A single oral dose of 400 mg moxifloxacin is included as a positive control in terms of the effect on cardiac repolarisation.

Study hypothesis:

Treatment with therapeutic (2 mg) or supratherapeutic (10 mg) doses of prucalopride in healthy male and female volunteers will not increase QTc interval compared to placebo.

DETAILED DESCRIPTION:
A total number of 120 healthy subjects (with an approximate 1:1 female:male ratio) are planned to be randomised.

Day 1: a baseline ECG profile. Day 1: Group 1 will receive prucalopride, Group 2a will receive moxifloxacin, and Group 2b will receive placebo.

On Day 5 (steady-state level is reached), a full ECG assessment day will be performed, enabling the comparison of prucalopride 2 mg with placebo.

Subsequently, the number of tablets will be escalated in all groups (blinded) with 1 tablet a day up to 5 tablets.

On Day 13 (steady state for the supratherapeutic dose level of 10 mg of prucalopride) another ECG assessment day will be performed, enabling a comparison of prucalopride 10 mg with placebo.

Group 2b will receive a single dose of moxifloxacin on Day 15. All subjects will be discharged on Day 16. Subjects will remain in the CRU throughout the treatment period.

All subjects will return for a follow-up visit on Day 30 (± 1 week) (approximately 14 days after the last dose).

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy volunteers aged between 18 to 50 years.
2. Body mass index (BMI) between 18 and 30 kg/m2.
3. Female subjects must:

   * be of childbearing potential with a negative serum β-human chorionic gonadotropin (β-HCG) test at screening, and be willing and able to use medically acceptable double barrier methods of birth control, throughout the whole study; or
   * be postmenopausal; or
   * have received surgical sterilisation at least 6 months before screening; AND
   * females must not be receiving hormone replacement therapy (HRT).

Main exclusion Criteria:

1. Abnormal QTcF and/or heart rate/blood pressure values at baseline.
2. Subjects with ECG abnormalities that may interfere with the accurate assessment of the QT interval.
3. Subjects with known cardiovascular disorders.
4. Subjects with known clinically significant arrhythmias.
5. Subjects with risk factors e.g., Torsades de Pointes.
6. Subjects with clinically relevant, abnormal serum electrolytes or complete blood count (CBC) at screening.
7. Female subjects who are lactating or pregnant.
8. Subjects suffering from other significant medical conditions.
9. Subjects with a known allergy or sensitivity to moxifloxacin, or to prucalopride.
10. Subjects with a positive screening test for hepatitis B, hepatitis C, or HIV at screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Treatment with therapeutic (2 mg) or supratherapeutic (10 mg) doses of prucalopride in healthy male and female volunteers does not increase QTc interval compared to placebo. | January to April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Remi VD Broeck, MD, Study Director — Movetis NV

REFERENCES:
- [Derived] Mendzelevski B, Ausma J, Chanter DO, Robinson P, Kerstens R, Vandeplassche L, Camm J. Assessment of the cardiac safety of prucalopride in healthy volunteers: a randomized, double-blind, placebo- and positive-controlled thorough QT study. Br J Clin Pharmacol. 2012 Feb;73(2):203-9. doi: 10.1111/j.1365-2125.2011.04088.x. PMID 21848574